CLINICAL TRIAL: NCT05733793
Title: A Retrospective-prospective, Multicenter, Observational Study Aimed to Record Molecular Data and to Explore Their Correlations With Clinical Outcomes in Gynecological Cancer Patients. The MITO GYNecological Cancers GEnetic Profile Registry (GYNGER) Study.
Brief Title: Molecular Data and Their Correlations With Clinical Outcomes in Gynecological Cancer Patients.
Acronym: GYNGER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Other Study IDs: Gynger
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Gynecologic Cancer
Keywords: Next Genaration Sequencing (NGS); Molecular profile

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort A (Retrospective):: Cohort A (Retrospective):
  • All consecutive patients diagnosed with gynecological malignancies who have performed an NGS analysis on tumor sample as for clinical practice or as part of a clinical study from the January 1st 2015 until the date in which the study is approved by the local ethical committee (Investigator is allowed to enroll patients) will be enrolled.
  Interventions: Other: NGS tests
- Cohort B (Prospective):: • All consecutive patients diagnosed with a gynecological malignancy who perform an NGS analysis on tumor sample as for clinical practice or as part of a clinical practice from the date in which the study is approved by the local ethical committee (Investigator is allowed to enroll patients) until 1st January 2025.
  Interventions: Other: NGS tests

INTERVENTIONS:
Other: NGS tests — This study is an observational, the patients with have an available NGS report performed in context of clinical practice or collected in clinical trials.
  Patients enrolled in the current study will be managed as for clinical practice and no additional genetic tests or other procedure will be required.

SUMMARY:
Gynger is a no profit, observational study, composed of a retrospective cohort (A) and a prospective cohort (B). The primary aim of this trial is to describe gene profile of Italian gynecological cancers patients, through the centralization of NGS reports performed in clinical practice or collected in clinical trials, and to correlation them with clinical and pathologic features.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form;
2. Female sex;
3. Age ≥18 years;
4. Diagnosis of a gynecological malignancy (ovarian cancer, uterine cancer, vulvar-vaginal cancer, gestational trophoblastic tumor);
5. Availability of NGS report performed on solid tumor tissue from primary or recurrent disease or liquid biopsy; data from NGS assays both in-house (academic test) and commercials can be used regardless of the number of genes analyzed

Exclusion Criteria:

* Patients for which the NGS analysis has been performed of germline tissue

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with a gynecological cancer with an available NGS report.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-06-16 (Actual); Primary Completion 2025-06-16 (Estimated); Study Completion 2025-06-16 (Estimated)

PRIMARY OUTCOMES:
The proportion of different gene alterations found with NGS tests | 4years
  This percentage will be calculated within enrolled patients that have a report of NGS test at baseline

SECONDARY OUTCOMES:
Progression-free-survival (PFS) | until progression disease (up to 4 years)
  PFS as defined by the Investigator using RECIST 1.1, as the time frame from randomization to progression or death for any cause,whichever comes first
Overall survival (OS) | 4 years
  Overall survival (OS) will be defined as the time between first line therapy start and death from any cause
ORR | 4 years
  Overall Response Rate (ORR) will be defined as the proportion of patients achieving a complete or partial response to a given therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Nazionale Tumori, IRCCS, Fondazione G Pascale, Naples, Italy

REFERENCES:
- See also: Description: Sponsor web-site for study conduction — https://usc.istitutotumori.na.it